CLINICAL TRIAL: NCT05124522
Title: Developing A Person-centered Internet-based Health Action Process Approach to Promoting Physical Activity in People With Multiple Sclerosis
Brief Title: A Health Action Process Approach Online Intervention for People With Multiple Sclerosis
Acronym: eHAPA-MS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Chung-Yi Chiu, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18754; RG-1706-27718 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2021-10-25; First posted 2021-11-18 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: Physical Activity; Internet-Based Intervention
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSPA eClass (Experimental)
  Interventions: Behavioral: MSPA eClass
- Waiting list (No Intervention)

INTERVENTIONS:
Behavioral: MSPA eClass — An 8-week MS-HAPA Internet-based intervention
  Arms: MSPA eClass

SUMMARY:
The purpose of this study is to implement the person-centered internet-based Health Action Process Approach to promoting physical activity in people with Multiple Sclerosis (i.e., eHAPA-MS online intervention) and assess the intervention's effectiveness and adherence.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years old and above;
* any type of multiple sclerosis
* have not maintained 30 minutes of MVPA accumulated per day for 2 days of the week during the previous 6 months;
* be relapse-free for the past 30 days;
* show low risk for contraindications of physical activity indicated by no more than a single 'yes' response on the Physical Activity Readiness Questionnaire;
* be able to walk with or without an assistive device;
* are willing to be randomized to an intervention or control group, complete the surveys and questionnaires, and wear an accelerometer during the intervention period;
* have a reliable Internet access.

Exclusion Criteria:

* have a score >14 for the leisure score index of the Godin Leisure-Time Exercise Questionnaire;
* No computer or mobile device access with the internet.
* Patient determined disease steps (PDDS) Score = 7 i.e., using a wheelchair or scooter most of the time, or PDDS Score = 8 being bedridden.
* Anyone living outside of the United States of America.
* Anyone who is unable to speak, read and write in English.
* not willing to be randomized to an intervention or control group, complete the surveys and questionnaires, and wear an accelerometer during the intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Health Action Process Approach Battery | Through study completion, an average of 1 month
  The battery measures risk perception, exercise benefits, motivation, and volition.
  "change" is being assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Chungyi Chiu, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (1):
- University of Illinois Urbana-Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The intervention result report.
Supporting Information: CSR
Time Frame: Anticipated December 2025

REFERENCES:
- [Derived] Chiu C, Sridharan V, Khaliji M, Sajib MRUZ, Gao X, Zackowski K. Patient-Centered, Theory-Based, Online Intervention to Promote a Physically Active Lifestyle for People With Multiple Sclerosis: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jul 17;14:e66091. doi: 10.2196/66091. PMID 40455827